CLINICAL TRIAL: NCT05866146
Title: A Pilot Randomized Control Trial to Test the Feasibility of Evaluating the Effectiveness of an Interprofessional Rehabilitation Program for Patients With Chronic Low Back Pain in Ethiopia: A Study Protocol
Brief Title: Feasibility of an Interprofessional Rehabilitation Program for Chronic Low Back Patients in the Ethiopian Health Setting
Acronym: IRP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Queen's University (Other)
Collaborators: MasterCard Foundation Scholarship Program (Unknown)
Responsible Party: Principal Investigator, Sintayehu Wami, Principal investigator, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ETH-IRP-CLBP-001; MCF (Other Grant/Funding Number: MasterCard Foundation Scholarship program)
Record Dates: First submitted 2023-04-18; First posted 2023-05-19 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Chronic Low-back Pain
Keywords: Low back pain; Multidisciplinary rehabilitation; Interprofessional rehabilitation; Biopsychosocial; Low back pain management
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: A two-arm parallel single-blinded pilot randomized control trial (RCT) will be employed to evaluate the feasibility and preliminary effectiveness of an interprofessional rehabilitation program compared to the usual care in patients with CLBP. Each eligible patient will have an equal chance to be allocated to the intervention or control group. Those who provide informed consent will complete a baseline assessment before being randomly assigned to the intervention or the control group without knowing the allocation of the group. Each group will be allocated/randomized 1:1 to the intervention and control groups. Except for the intervention being evaluated, all groups will be treated identically in every way.
Who Masked: Outcomes Assessor
Masking Description: In this study, research staff collecting outcome data from patients will be blinded to the group allocation. However, the treating health professionals and patients will not be blinded to group allocation due to the nature of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interprofessional rehabilitation program (Experimental): Participants of the intervention group will receive an interprofessional rehabilitation program, which involve a combination of physical, psychological, behavioral, and/or vocational components, for four weeks.
  Interventions: Other: Interprofessional rehabilitation program
- Usual standard care (Active Comparator): The control group participants will receive the usual standard care according to the current practices at the University of Gondar specialized hospital over the same four weeks.
  Interventions: Other: Usual standard care

INTERVENTIONS:
Other: Interprofessional rehabilitation program — The interprofessional rehabilitation program includes a comprehensive assessment, intensified physical activities and exercises, pain education, psychotherapy, occupational therapy, ergonomic interventions, and psychosocial counselling in addition to the current treatment standards. The interprofessional rehabilitation program will be delivered in a combination of individual (one-to-one) and group sessions (in groups of 6 - 10 patients). Care providers will apply a combination of lectures and discussions, individual exercises, and group-based exercises and education. All sessions will be delivered face-to-face (in person). The intervention will be provided by a team of healthcare providers with different professional backgrounds and training. The interprofessional team may include experienced physicians (GPs), neurosurgeons, physiotherapists, nurses, occupational therapists, and clinical psychologists.
  Other Names: Multidisciplinary rehabilitation program
  Arms: Interprofessional rehabilitation program
Other: Usual standard care — Participants in this group will receive the usual care currently implemented mainly pharmacological treatment (pain medication), and back pain advice. The usual care in rare occasions may also include physical therapy such as exercise and massage.
  Other Names: Routine care
  Arms: Usual standard care

SUMMARY:
The overall aim of this pilot RCT is to assess the feasibility of conducting a future definitive randomized control trial (RCT) for evaluating the effectiveness of an interprofessional rehabilitation program compared to the usual care in adults with chronic low back pain in Ethiopia.

Specific objectives of this study include:

* To evaluate the feasibility of trial procedures (recruitment rate, retention rate, adherence rate).
* To explore the feasibility and acceptability of the intervention from the patients' and care providers' perspectives.
* To estimate the preliminary treatment effect and standard deviation of the relevant clinical outcome measures (physical functioning, pain intensity, workability, HRQoL, psychological functioning) in patients with CLBP to inform sample size calculation for the definitive RCT.

Patients with chronic low back pain diagnosed through focused history and physical examination are accepted for enrolment. Each eligible patient will have an equal chance to be allocated to the intervention or control group.

Participants of the intervention group will receive interprofessional rehabilitation for four weeks. Participants of the intervention group will receive interprofessional rehabilitation that contain components aimed at enabling optimal physical, psychological, and social functioning, including addressing the work abilities of patients. The components will include a comprehensive assessment, intensified physical activities and exercises, pain education, psychological support, occupational therapy, ergonomic interventions, and vocational counselling.

Participants in the comparison group will receive the usual care according to the current standard care for patients with chronic low back pain at the University of Gondar specialized referral hospital in Ethiopia for over four weeks.

DETAILED DESCRIPTION:
Chronic low back pain (CLBP) is the most common type of musculoskeletal pain, and it has a substantial negative consequence on the ability to engage in meaningful activities, participation in work, health-related quality of life, and social relationships. CLBP-related disability is increasing worldwide, and the majority of this increase is associated with the growing burden in low-and-middle-income countries, including Ethiopia.

A growing body of evidence from high-income countries indicates the effectiveness of interprofessional rehabilitation programs for patients with CLBP. The currently implemented biomedically focused fragmented care in low- and middle-income countries appears to have limited lasting effect, owing to long-term disability. Therefore, this pilot RCT aims to evaluate the feasibility of conducting a definitive RCT to assess the effectiveness of an interprofessional rehabilitation program compared to the usual care for patients with CLBP in Ethiopia. Accordingly, the investigators will evaluate some elements of full RCT, including recruitment and retention rate, adherence, acceptability of the intervention, sample size estimation, and participants' preliminary responses to the interventions. Hence, this study will substantially benefit in informing components of the main trial design, minimizing uncertainties, and increasing the likelihood of successfully conducting the definitive RCT in the future. In addition, this pilot RCT is expected to provide a source of evidence for other initiatives aimed at developing and implementing interprofessional rehabilitation programs in a similar context.

A two-arm parallel single-blinded pilot randomized control trial (RCT), with embedded qualitative interviews, will be employed to assess the feasibility of conducting a full RCT to evaluate the effectiveness of an interprofessional rehabilitation program compared to the usual care in patients with CLBP.

Sample size: The investigators will recruit a total of 40 (i.e., 20 in the intervention group and 20 in the control group) patients with CLBP.

A simple block randomization method with random block sizes of 4 to 8 will be employed to randomize participants into the intervention and control groups.

Data collection procedures: The data will be collected by a trained research assistant who will be blind to the group assignment using interviewer administered approach at three time points: at baseline before the start of the intervention, the 5th week immediately following the final visit for the intervention, and the 16th week (after 12 weeks of intervention completion) to investigate whether the effects are sustained over time after the completion of the intervention.

In addition to the primary and secondary outcome measures, the study participants' socio-demographic and behavioural characteristics, such as age, sex, educational level, marital status, and physical activities, will be collected at the baseline. A two-day training will be given to data collectors about the trial process, outcome measures, and tools used by PI.

For the embedded qualitative interviews, a research assistant will conduct a face-to-face, in-depth interview with treating health professionals and study participants during the intervention phase. A semi-structured interview guide will be used to conduct an interview. The interview will be conducted to explore the acceptability of the intervention and barriers and facilitators associated with the implementation of the intervention from both treating health professionals' and participants' perspectives. The investigators will also explore the perceptions and experiences of the study participants about the intervention they have received.

Data management and statistical analysis: Descriptive statistics like mean, standard deviation, proportions, and frequency distributions of all variables will be computed. The quantitative data analysis will be performed using SPSS version 27. The main analysis will be performed according to the intention-to-treat (ITT) principle.

The thematic text analysis approach as described by Braun and Clarke will be used to analyze the qualitative data.

ELIGIBILITY:
Inclusion Criteria:

* Adults above the age of 18 years
* Patients with chronic low back pain ('pain and discomfort localized below the costal margin and above the inferior gluteal folds, with or without leg pain') that persists for 3 months or more will be included in this trial

Exclusion Criteria:

* Patients who have serious known spinal pathology (e.g., tumours, vertebral fractures, and inflammatory diseases), and spinal surgery within the last 12 months will be excluded.
* Participants with CLBP due to specific pathologies (e.g., infections, neoplasms, metastases, fractures, osteoporosis, rheumatoid arthritis, radiculopathies) or other inflammatory articular conditions (for example, ankylosing spondylitis), spinal stenosis, or fracture will also be excluded from the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-05-20 (Estimated); Primary Completion 2023-07-15 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Patient recruitment rate | The data will be collected at the baseline before the start of the intervention.
  The recruitment rate is described as the number of eligible patients with CLBP recruited and randomized within two to three months at the University of Gondar specialized hospital. Hence, the recruitment rate will be calculated by dividing the total number of patients with CLBP recruited at the University of Gondar specialized hospital by the total recruitment period (number of months).
Patient retention rate | The data will be collected through intervention completion, up to five weeks.
  The number of patients recruited, randomized, and considered for the analysis will be used to calculate the retention rate. The retention rate will be calculated as the percentage of participants that complete all secondary outcome measures.
Intervention adherence rate | The data will be collected through intervention completion, up to five weeks.
  The intervention adherence rate will be determined by calculating the proportion of group and individual intervention sessions completed by the study participants as per the stated intervention protocol.
Acceptability of intervention and trial procedures | The data will be collected through intervention completion, up to five weeks.
  A qualitative description approach will be employed to explore the acceptability of the intervention and trial procedures from both treating health professionals and study participants' perspectives through an in-depth interview using a semi-structured interview guide. intervention from the patients' and care providers perspectives.
Treatment fidelity | The data will be collected through intervention completion, up to five weeks.
  The investigators will evaluate whether the intervention is delivered with fidelity according to the developed protocol. The care providers will assess and rate using a treatment fidelity checklist at each visit to evaluate treatment fidelity. Fidelity will be judged acceptable if the score is > 80% compatible with the intervention protocol.

SECONDARY OUTCOMES:
Physical functioning | At baseline before the start of the intervention, the 5th week , and the 16th week (after 12 weeks of intervention completion).
  The cross-culturally adapted and validated Roland Morris Disability Questionnaire (RMDQ-24) will be used to measure the physical functioning of patients with CLBP. The RMQ is a 24-item patient-reported outcome measure that inquires about pain-related disability resulting from LBP. Each item is given a 1 (Yes) or 0 (No) score ranging from 0 to 24; higher scores represent higher levels of pain-related disability.
Pain intensity | At baseline before the start of the intervention, the 5th week , and the 16th week (after 12 weeks of intervention completion).
  Pain intensity will be measured using a brief pain inventory - short form (BPI-sf) standard questionnaire. The Brief Pain Inventory - Short Form (BPI-sf) is a nine-item self-administered questionnaire that is used to assess the degree of a patient's pain and its influence on daily functioning. On a 10-point scale, the patient is asked to rate their worst, least, average, and current pain intensity. A score of 1 - 4 = Mild Pain, 5 - 6 = Moderate Pain and a score of 7 - 10 = Severe Pain.
Health-related quality of life | At baseline before the start of the intervention, the 5th week , and the 16th week (after 12 weeks of intervention completion).
  Will be measured using the 36-item short-form health survey (SF-36) questionnaire. Possible scores range from 0 to 100, with higher scores representing better health status.
Self-efficacy | At baseline before the start of the intervention, the 5th week , and the 16th week (after 12 weeks of intervention completion).
  To measure self-efficacy of patients with CLBP, the investigators will utilize the pain self-efficacy questionnaire (PSEQ). The PSEQ is a ten-item questionnaire in which patients assess their level of confidence on a scale of 0 (not at all confident) to 6 (very confident) (completely confident). Total scores are derived by adding the individual items' values, which range from 0 (low self-efficacy) to 60 (high self-efficacy) (more self-efficacy).
Global rating of change | At baseline before the start of the intervention, the 5th week , and the 16th week (after 12 weeks of intervention completion).
  The Global Rating of Change (GRC) scales are used to assess self-perceived improvement/changes in health. To measure the global rating of change, the investigators will use an 11-point global rating of change scale (GROC) (-5 to +5), ranging from -5 (very much worse), through 0 (unchanged) to +5 (completely recovered).
Psychological functioning | At baseline before the start of the intervention, the 5th week , and the 16th week (after 12 weeks of intervention completion).
  The investigators will use the Hospital Anxiety and Depression Scale (HADS) to measure psychological functioning. Scoring for each item ranges from zero to three, with three denoting the highest anxiety or depression level. A total subscale score of >8 points out of a possible 21 denotes considerable symptoms of anxiety or depression.

CONTACTS AND LOCATIONS:
Overall Officials: Sintayehu Da Wami, Principal Investigator — Queen's University

IPD SHARING:
Plan to Share IPD: No
Efforts will be made to present the results at scientific conferences and publish them in a peer-reviewed journal.